CLINICAL TRIAL: NCT07089251
Title: The Perioperative Outcome of Epinephrine Infusion and Tranexamic Acid in Knee Arthroplasty Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Wazzan Saleh ALJuhani, Principal investigator, Orthopedic Surgeon, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICTR24/002/9
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Knee Arthroplasty, Total; Knee Arthritis, Osteoarthritis; Total Knee Anthroplasty; Blood Loss; Tranexamic Acid Use; Epinephrine
MeSH Terms: conditions — Osteoarthritis; Hemorrhage | interventions — Epinephrine; Tranexamic Acid; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine + Tranexamic Acid Group (Experimental): The experimental group will receive both epinephrine and tranexamic acid
  Interventions: Drug: low-dose epinephrine and tranexamic acid
- Tranexamic Acid Group (Active Comparator): The comparator group will receive only tranexamic acid
  Interventions: Drug: Tranexamic Acid (TXA) treatment

INTERVENTIONS:
Drug: low-dose epinephrine and tranexamic acid — low-dose epinephrine and tranexamic acid
  Arms: Epinephrine + Tranexamic Acid Group
Drug: Tranexamic Acid (TXA) treatment — Tranexamic Acid
  Arms: Tranexamic Acid Group

SUMMARY:
The aim of this clinical trial is to evaluate the effect of administering low-dose epinephrine and tranexamic acid on perioperative blood loss, thromboembolic complications, and hospitalization duration in patients undergoing knee joint arthroplasty.

Also aim to evaluate the effect of administering low-dose epinephrine and tranexamic acid on perioperative thromboembolic complications, and hospitalization duration

DETAILED DESCRIPTION:
Patients will be randomly divided into two groups: one receiving intravenous low-dose epinephrine and tranexamic acid, while the other will receive TXA alone as the control. Randomization to be done using a computer-generated table.

The study will be done a superiority clinical trial. with an estimated 24 hour blood loss of 300 ml, with standard deviation of 150 ml. a power of 80% and alpha 5%, an estimated sample size of 80 is needed to detect a difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing knee joint arthroplasty.
* Saudi and Non-Saudi Patient.
* Patients who have Complete medical record.

Exclusion Criteria:

* End stage renal disease
* Liver cirrhosis
* Coagulopathy
* Pre-operative Hgb <10 5.
* History of cerebrovascular accident or myocardial infarction in past 12 months.
* History of Heart failure.
* History of arrhythmia.
* History of pheochromocytoma, thyrotoxicosis and glaucoma.
* Pregnancy or breast feeding
* History of Deep venous thrombosis or pulmonary embolism
* Allergy to epinephrine or tranexamic acid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood loss | Daily, till post-operative day 5
  Calculated 24 h blood loss in mL, Hidden blood loss in mL, Hemoglobin levels in g/dL, Hematocrit levels as a percentage, Platelets count in cells/µL.

SECONDARY OUTCOMES:
Thromboembolic complications | Daily, till post-operative day 5
Hospitalization duration | Daily, till post-operative day 5
Drug side effects (epinephrine + tranexamic acid) | Daily, till post-operative day 5
Complications | Daily, till post-operative day 5
  VTE, SSI, UTI, AKI, Cardiac Arrhythmias, Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Wazzan Aljuhani, MD, FRCSC, MBA, MMEd, Principal Investigator — King Abdulaziz Medical City, MNGHA
Locations (1):
- King Abdulaziz Medical City, Ministry of National Guard - Health Affairs, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes